CLINICAL TRIAL: NCT04437082
Title: Performance Evaluation of OCT and OCTA-based Ocular Measurements
Brief Title: Performance Evaluation of OCT and OCT Angiography-based Ocular Measurements (Optical Coherence Tomography)
Acronym: OCT
Status: Completed | Type: Observational
Sponsor: Optovue (Industry)
Responsible Party: Sponsor
Other Study IDs: 200-54611
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-02

CONDITIONS: Normal Eyes and Ocular Pathology
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Normal: no pre-existing conditions
  Interventions: Device: optical coherence tomography
- Glaucoma: diagnosis of glaucoma
  Interventions: Device: optical coherence tomography
- Retina: diagnosis of retina pathology
  Interventions: Device: optical coherence tomography
- Cornea: diagnosis of corneal condition
  Interventions: Device: optical coherence tomography

INTERVENTIONS:
Device: optical coherence tomography — imaging structural and vascular features of the eye

SUMMARY:
The purpose of this study is to assess performance of measurements of anatomical and vascular structures of the eye based on OCT and OCTA scans in normal subjects and eyes with pathology.

ELIGIBILITY:
Inclusion Criteria:

* Normal - No pre-existing conditions.
* Glaucoma - Diagnosis of glaucoma.
* Retina - Diagnosis of retinal pathology
* Cornea - Diagnosis of clinic condition.

Exclusion Criteria:

- Unable to complete required exams.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Seeing eye doctor for routine or follow-up care
Sampling Method: Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Standard Deviation | Day 1
  measure of variance

CONTACTS AND LOCATIONS:
Locations (1):
- Oklahoma College of Optometry, Northeastern State University, Tahlequah, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No